CLINICAL TRIAL: NCT03136185
Title: A Multi-Center, Open Label Study to Assess the Safety, Steady-State Pharmacokinetics and Pharmacodynamics of IMG-7289 in Patients With Myelofibrosis
Brief Title: Bomedemstat (IMG-7289/MK-3543) in Participants With Myelofibrosis (IMG-7289-CTP-102/MK-3543-002)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMG-7289-CTP-102; IMG-7289-CTP-102 (Other: Imagobio); MK-3543-002 (Other: Merck); 2018-003811-23 (EudraCT Number)
Record Dates: First submitted 2017-04-18; First posted 2017-05-02 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Myelofibrosis; Post-polycythemia Vera Myelofibrosis (PPV-MF); Post-essential Thrombocythemia Myelofibrosis (PET-MF); Primary Myelofibrosis (PMF)
Keywords: LSD1
MeSH Terms: conditions — Primary Myelofibrosis | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d (Experimental): In the Phase 1/2a portion of the study, PMF participants received 0.25 mg/kg/d bomedemstat orally every day (qd) for 85 days during the Initial Treatment Period (ITP). Qualifying participants could continue to receive treatment for an additional 85 days during an Additional Treatment Period (ATP) as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d (Experimental): In the Phase 1/2a portion of the study, PPV-MF participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 85 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d (Experimental): In the Phase 1/2a portion of the study, PET-MF participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 85 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PMF: Bomedemstat 0.5 mg/kg/d (Experimental): In the Phase 2b portion of the study, PMF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d (Experimental): In the Phase 2b portion of the study, PPV-MF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d (Experimental): In the Phase 2b portion of the study, PET-MF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PMF: Bomedemstat 0.6 mg/kg/d (Experimental): In the Phase 2b portion of the study, PMF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d (Experimental): In the Phase 2b portion of the study, PPV-MF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat
- Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d (Experimental): In the Phase 2b portion of the study, PET-MF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during an ATP as determined by the investigator. The ATP could repeat indefinitely in participants that continued to derive clinical benefit.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Oral (capsule) administration according to dose allocation.
  Other Names: IMG-7289; MK-3543; LSD1 inhibitor

SUMMARY:
This is a Phase 1/2 open-label study to evaluate the safety, tolerability, steady-state pharmacokinetic (PK) and pharmacodynamics (PD) of a lysine-specific demethylase 1 (LSD1) inhibitor, bomedemstat (IMG-7289/MK-3543), administered orally once daily in participants with myelofibrosis.

The primary hypothesis is that bomedemstat is a safe and tolerable orally available agent when administered to participants with myelofibrosis including primary myelofibrosis (PMF), post-polycythaemia vera-myelofibrosis (PPVMF), and post-essential thrombocythaemia-myelofibrosis (PET-MF) (collectively referred to as 'MF'); inhibition of LSD1 by bomedemstat will reduce spleen size in those with splenomegaly, improve haematopoiesis and reduce constitutional symptoms associated with these disorders.

DETAILED DESCRIPTION:
This study initiated as a Phase 1/2a study assessing the safety of the starting dose, an 85-day duration of treatment, and the PK and PD effects of bomedemstat, with transition to a Phase 2b study incorporating changes supported by the Phase 1/2a data.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of either PMF per World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms, or PPV-MF or PET-MF per the International Working Group for Myelofibrosis Research and Treatment
* High or intermediate-2 risk disease

Exclusion Criteria:

* Receiving other treatments for the condition (with exceptions and time limits)
* Major surgery in last 4 weeks, any surgery in the last 2 weeks
* History of, or scheduled, hematopoietic stem cell transplant within 24 weeks of Screening
* History of splenectomy
* Current use of prohibited medications
* A concurrent second active and nonstable malignancy
* Known human immunodeficiency virus infection or active Hepatitis B or Hepatitis C virus infection
* Other hematologic/biochemistry requirements, as per protocol
* Use of an investigational agent within last 14 days
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- University of Michigan, Ann Arbor, Michigan, United States
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Universitatsklinikum Essen, Essen, Germany
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy
- Guy's and St Thomas' Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PPV-MF), and post-essential thrombocythemia myelofibrosis (PET-MF) were recruited for this study.
Pre-assignment Details: Eighteen participants were enrolled in the Phase 1/2a portion of this study and 72 participants were enrolled in the Phase 2b portion of this study.
Groups:
- Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d: In the Phase 1/2a portion of the study, PMF participants received 0.25 mg/kg/d bomedemstat orally every day (qd) for 85 days during the Initial Treatment Period (ITP). Qualifying participants could continue to receive treatment for an additional 169 days during the Additional Treatment Period (ATP) as determined by the investigator.
- Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d: In the Phase 1/2a portion of the study, PPV-MF participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d: In the Phase 1/2a portion of the study, PET-MF participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PMF: Bomedemstat 0.5 mg/kg/d: In the Phase 2b portion of the study, PMF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d: In the Phase 2b portion of the study, PPV-MF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d: In the Phase 2b portion of the study, PET-MF participants received 0.5 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PMF: Bomedemstat 0.6 mg/kg/d: In the Phase 2b portion of the study, PMF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d: In the Phase 2b portion of the study, PPV-MF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d: In the Phase 2b portion of the study, PET-MF participants received 0.6 mg/kg/d bomedemstat orally qd for 169 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
Period: Overall Study
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Started | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Treated | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Entered Additional Treatment Period (ATP) | 6 | 2 | 3 | 3 | 1 | 4 | 17 | 5 | 9
Completed Initial Treatment Period (ITP) | 7 | 3 | 4 | 4 | 1 | 4 | 18 | 8 | 10
Completed | 1 | 0 | 0 | 2 | 0 | 3 | 14 | 5 | 7
Not Completed | 8 | 3 | 6 | 6 | 5 | 8 | 10 | 6 | 6
Not completed — Adverse Event | 0 | 1 | 3 | 1 | 2 | 2 | 5 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 1
Not completed — Protocol Defined Disease Progression | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 3
Not completed — Not Reported | 4 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d: In the Phase 1/2a portion of the study, PMF participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
- Total: Total of all reporting groups
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d | Total
Number analyzed (Participants) | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (12.43) | 74.7 (5.51) | 64.7 (6.59) | 69.6 (8.38) | 64.8 (7.46) | 69.4 (14.40) | 65.2 (9.42) | 66.7 (9.27) | 61.3 (12.07) | 65.7 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 4 | 4 | 6 | 12 | 8 | 4 | 43
  Male | 8 | 3 | 2 | 4 | 1 | 5 | 12 | 3 | 9 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 8 | 3 | 5 | 8 | 4 | 10 | 22 | 11 | 9 | 80
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 5 | 5 | 21
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 7 | 2 | 6 | 7 | 4 | 9 | 12 | 6 | 6 | 59
  Other | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Reported | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any one of the following adverse events (AEs) that occured through Day 7 of the Initial Treatment Period (ITP) and was considered by the Investigator to be possibly, probably or definitely related to bomedemstat:
  * Thrombocytopenia leading to clinically significant sequelae (i.e., a clinically significant bleeding event or the need for prophylactic transfusions)
  * A clinically significant bleeding event in a participant with a platelet count >50 x 10^9/L (50 k/μL)
  * Any Grade 4 or 5 non-haematologic adverse event
  * Any Grade 3 non-haematologic adverse event with failure to recover to Grade 2 within 7 days of drug cessation, with the following exceptions: ≥ Grade 3 nausea, vomiting or diarrhea that responds to standard medical care; ≥ Grade 3 aesthenia lasting less than 14 days; any Grade 3 electrolyte abnormality unrelated to the underlying malignancy and persisting greater than 24 hours.
  The number of participants with a DLT were reported.
Time Frame: Up to Day 7 of the ITP
Population: All participants receiving at least one dose of bomedemstat were included in the DLT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: An AE was any undesirable physical, psychological or behavioral effect experienced by a participant, in conjunction with the use of the drug or biologic, whether or not product-related. This included any untoward signs or symptoms experienced by the participant from the time of first dose with bomedemstat until completion of the study. Serious AEs (SAEs) were any AE that resulted in death, life-threatening experience, required or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly, or important medical events. The number of participants with at least one treatment-emergent (TE) SAE was reported for each arm.
Time Frame: Up to approximately 30 months
Population: All participants receiving at least one dose of bomedemstat were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Participants | 4 | 2 | 5 | 4 | 4 | 7 | 12 | 3 | 3

3. Primary Outcome: Number of Participants With Adverse Events
Description: An AE was any undesirable physical, psychological or behavioral effect experienced by a participant, in conjunction with the use of the drug or biologic, whether or not product-related. This included any untoward signs or symptoms experienced by the participant from the time of first dose with bomedemstat until completion of the study. The number of participants with at least one TE AE was reported for each arm.
Time Frame: Up to approximately 30 months
Population: All participants receiving at least one dose of bomedemstat were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Participants | 9 | 3 | 6 | 8 | 5 | 11 | 23 | 10 | 12

4. Primary Outcome: Number of Participants That Discontinued Study Treatment Due To AEs
Description: An AE was any undesirable physical, psychological or behavioral effect experienced by a participant, in conjunction with the use of the drug or biologic, whether or not product-related. This included any untoward signs or symptoms experienced by the participant from the time of first dose with bomedemstat until completion of the study. The number of participants that discontinued study treatment with bomedemstat due to a TE AE was reported for each arm.
Time Frame: Up to approximately 29 months
Population: All participants receiving at least one dose of bomedemstat were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 9 | 3 | 6 | 8 | 5 | 11 | 24 | 11 | 13
Participants | 0 | 1 | 5 | 1 | 2 | 4 | 5 | 2 | 3

5. Primary Outcome: Phase 1/2a Portion: Observed Maximum Concentration (Cmax) of Bomedemstat
Description: Cmax was defined as the maximum observed concentration after administration obtained directly from the concentration time profile. Blood and plasma samples were collected at pre-specified timepoints to calculate Cmax in participants of the Phase 1/2a portion of the study. As pre-specified by the protocol and Pharmacokinetic Analysis Plan (PAP), Phase 2b participants were excluded from this analysis.
Time Frame: Day 21: Pre-dose and 0.5, 1, 2, 3, 4, 8, and 24 hours (Day 22) after dosing.
Population: As pre-specified by the PAP, all participants in the Phase 1/2a portion of the study who received bomedemstat and completed a sufficient portion of the study with enough data for the determination of pharmacokinetic parameters were analyzed. For the purposes of the analysis, Phase 1/2a participants were analyzed irrespective of myelofibrosis disorder (PMF, PPV-MF, or PET-MF) per protocol. Phase 2b participants were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Ph 1/2a Portion: Bomedemstat 0.25 mg/kg/d: In the Phase 1/2a portion of the study, participants received 0.25 mg/kg/d bomedemstat orally qd for 85 days during the ITP. Qualifying participants could continue to receive treatment for an additional 169 days during the ATP as determined by the investigator.
Arm/Group | Ph 1/2a Portion: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0 | 0
ng/mL
  Plasma | 12.63 (104.41) |  |  |  |  |  |
  Blood: number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0
  Blood | 26.27 (66.76) |  |  |  |  |  |

6. Primary Outcome: Phase 1/2a Portion: Time to Maximum Concentration (Tmax) of Bomedemstat
Description: Tmax was defined as the time to maximum concentration after administration obtained by inspection. Blood and plasma samples were collected at pre-specified timepoints to calculate Tmax in participants of the Phase 1/2a portion of the study. As pre-specified by the protocol and Pharmacokinetic Analysis Plan (PAP), Phase 2b participants were excluded from this analysis.
Time Frame: Day 21: Pre-dose and 0.5, 1, 2, 3, 4, 8, and 24 hours (Day 22) after dosing.
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Ph 1/2a Portion: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0 | 0
hour
  Plasma | 1.00 [0.50 to 2.85] |  |  |  |  |  |
  Blood: number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0
  Blood | 1.05 [0.50 to 3.02] |  |  |  |  |  |

7. Primary Outcome: Phase 1/2a Portion: Area Under the Concentration-time Curve of Bomedemstat From Time 0 to 24 Hours Post-dose (AUC0-24)
Description: AUC0-24 was defined as the area under the concentration versus time curve calculated using the linear trapezoidal rule from the zero time-point to the 24-hour time-point concentration. Blood and plasma samples were collected at pre-specified timepoints to calculate AUC0-24 in participants of the Phase 1/2a portion of the study. As pre-specified by the protocol and Pharmacokinetic Analysis Plan (PAP), Phase 2b participants were excluded from this analysis.
Time Frame: Day 21: Pre-dose and 0.5, 1, 2, 3, 4, 8, and 24 hours (Day 22) after dosing.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour•ng/mL
Arm/Group | Ph 1/2a Portion: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0 | 0
hour•ng/mL
  Plasma | 63.90 (68.56) |  |  |  |  |  |
  Blood: number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0
  Blood | 265.92 (68.92) |  |  |  |  |  |

8. Primary Outcome: Phase 1/2a Portion: Apparent Total Clearance (CL/F) of Bomedemstat After Oral Administration
Description: CL/F was defined as the apparent total clearance of drug after oral administration. Blood and plasma samples were collected at pre-specified timepoints to calculate CL/F in participants of the Phase 1/2a portion of the study. As pre-specified by the protocol and Pharmacokinetic Analysis Plan (PAP), Phase 2b participants were excluded from this analysis.
Time Frame: Day 21: Pre-dose and 0.5, 1, 2, 3, 4, 8, and 24 hours (Day 22) after dosing.
Population: As pre-specified by the PAP, only participants in the Phase 1/2a portion of the study who received bomedemstat and completed a sufficient portion of the study with enough data for the determination of pharmacokinetic parameters were analyzed. For the purposes of the analysis, Phase 1/2a participants were analyzed irrespective of myelofibrosis disorder (PMF, PPV-MF, or PET-MF) per protocol. Phase 2b participants were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Ph 1/2a Portion: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0 | 0
mL/min
  Plasma | 12787.43 (63.72) |  |  |  |  |  |
  Blood: number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0
  Blood | 3067.57 (85.78) |  |  |  |  |  |

9. Primary Outcome: Percentage Change From Baseline in Spleen Volume
Description: Change in spleen volume was assessed based on calculated spleen volume (ml) measured by magnetic resonance imaging (MRI), or computerized tomography (CT) scan (where locally permitted) if the participant was not a candidate for MRI from Day 0. Percentage change from baseline in spleen volume was reported at Initial Treatment Period (ITP) Day 84, ITP Day 168, Additional Treatment Period 1 (ATP1) Day 84 (Study Day 253), and ATP1 Day 168 (Study Day 337).
Time Frame: Baseline, ITP Day 84 (Study Day 84), ITP Day 168 (Study Day 168), ATP1 Day 84 (Study Day 253), and ATP1 Day 168 (Study Day 337)
Population: All allocated participants who received at least one dose of treatment and had available spleen volume data.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 3 | 6 | 17 | 8 | 8
Percentage Change
  ITP Day 84 (Study Day 84) | 3.3 [-50.5 to 57.0] | -13.7 [-49.6 to 22.2] | 2.2 [-110.3 to 114.8] | -9.1 [-27.9 to 9.6] | -7.2 [-80.2 to 65.8] | 0.3 [-32.3 to 32.9] | 10.0 [1.2 to 18.8] | -2.3 [-31.5 to 26.9] | 1.2 [-10.9 to 13.2]
  ITP Day 168 (Study Day 168): number analyzed (Participants) | 0 | 0 | 0 | 3 | 1 | 2 | 16 | 5 | 8
  ITP Day 168 (Study Day 168) |  |  |  | -23.9 [-43.2 to -4.6] | -19.6 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. | -33.7 [-43.8 to -23.6] | 12.3 [-4.1 to 28.6] | -15.4 [-56.7 to 25.8] | -4.4 [-20.6 to 11.8]
  ATP1 Day 84 (Study Day 253): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ATP1 Day 84 (Study Day 253) |  |  |  |  |  | -27.7 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  |  |
  ATP1 Day 168 (Study Day 337): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 2 | 5
  ATP1 Day 168 (Study Day 337) |  |  |  | -36.5 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  | -38.9 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. | 37.4 [-55.6 to 130.5] | 6.0 [-302.0 to 313.9] | -15.0 [-39.0 to 9.0]

10. Primary Outcome: Percentage Change From Baseline in Spleen Size
Description: Change in spleen size was assessed based on spleen palpation (in cm) at each visit. Percentage change from baseline in spleen size was reported at ITP Day 84, ITP Day 168, ATP1 Day 84 (Study Day 253), ATP1 Day 168 (Study Day 337), ATP2 Day 84 (Study Day 422), ATP2 Day 168 (Study Day 506), and ATP3 Day 84 (Study Day 591). As prespecified by the Statistical Analysis Plan, assessments for the Phase 1/2 groups were summarized using visit windowing after the Day 84 visit of the ITP to allow for comparison with the Phase 2b groups at ITP Day 168.
Time Frame: Baseline, ITP Day 84 (Study Day 84), ITP Day 168 (Study Day 168), ATP1 Day 84 (Study Day 253), ATP1 Day 168 (Study Day 337), ATP2 Day 84 (Study Day 422), ATP2 Day 168 (Study Day 506), and ATP3 Day 84 (Study Day 591)
Population: All allocated participants who received at least one dose of treatment and had available spleen size data.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 2 | 6 | 13 | 6 | 5
Percentage Change
  ITP Day 84 (Study Day 84): number analyzed (Participants) | 6 | 3 | 4 | 3 | 2 | 6 | 13 | 6 | 4
  ITP Day 84 (Study Day 84) | -36.5 [-68.0 to -5.0] | 9.6 [-95.1 to 114.2] | 24.1 [-79.4 to 127.7] | 20.7 [-132.2 to 173.7] | -28.1 [-257.8 to 201.6] | 11.0 [-70.7 to 92.7] | -34.7 [-58.1 to -11.3] | -38.2 [-53.4 to -23.1] | -59.6 [-113.4 to -5.7]
  ITP Day 168 (Study Day 168): number analyzed (Participants) | 4 | 1 | 2 | 1 | 0 | 2 | 11 | 6 | 4
  ITP Day 168 (Study Day 168) | -20.7 [-48.3 to 6.9] | -39.6 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. | 116.3 [-1794.8 to 2027.4] | -27.8 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  | -36.1 [-212.6 to 140.4] | -24.8 [-74.2 to 24.5] | -28.5 [-60.1 to 3.0] | -41.2 [-102.9 to 20.6]
  ATP1 Day 84 (Study Day 253): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 2 | 8 | 3 | 5
  ATP1 Day 84 (Study Day 253) |  |  |  | -27.8 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  | -36.1 [-212.6 to 140.4] | -27.9 [-84.8 to 29.0] | -50.4 [-101.7 to 0.9] | -28.4 [-97.7 to 40.9]
  ATP1 Day 168 (Study Day 337): number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 4
  ATP1 Day 168 (Study Day 337) | -19.0 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  |  | -27.8 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  | -38.9 [-180.1 to 102.3] | -1.9 [-151.0 to 147.3] | -38.9 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. | -82.4 [-117.4 to -47.4]
  ATP2 Day 84 (Study Day 422): number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  ATP2 Day 84 (Study Day 422) | -4.8 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  |  |  |  | -37.5 [-196.3 to 121.3] |  | -44.4 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |
  ATP2 Day 168 (Study Day 506): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ATP2 Day 168 (Study Day 506) |  |  |  |  |  | -22.0 [NA to NA] — 95% confidence intervals could not be calculated for arms with n<2 participants. |  |  |
  ATP3 Day 84 (Study Day 591): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  ATP3 Day 84 (Study Day 591) |  |  |  |  |  | -11.1 [-152.3 to 130.1] |  |  |

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: All-Cause Mortality table includes all allocated participants. Serious and Non-serious adverse events (AEs) tables include all allocated participants who received at least 1 dose of study drug.
Arm/Group | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/6 | 1/8 | 1/5 | 0/11 | 1/24 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 4/9 | 2/3 | 5/6 | 4/8 | 4/5 | 7/11 | 12/24 | 3/11 | 3/13
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 6/6 | 8/8 | 5/5 | 11/11 | 23/24 | 10/11 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d (N=9) | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d (N=3) | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d (N=6) | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d (N=8) | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d (N=5) | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d (N=11) | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d (N=24) | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d (N=11) | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 3 (8) | 2 (20) | 2 (2) | 5 (26) | 2 (2) | 2 (3) | 2 (6)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (6) | 1 (2) | 3 (17) | 4 (26) | 2 (5) | 7 (25) | 1 (2) | 3 (13) | 3 (7)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 1 (4) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 1 (1) | 2 (2) | 4 (7) | 1 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1) | 3 (5) | 0 (0) | 2 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (4) | 0 (0) | 1 (1) | 4 (10) | 2 (2) | 1 (1) | 1 (1) | 1 (4) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (6) | 1 (6) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ph 1/2a PMF: Bomedemstat 0.25 mg/kg/d (N=9) | Ph 1/2a PPV-MF: Bomedemstat 0.25 mg/kg/d (N=3) | Ph 1/2a PET-MF: Bomedemstat 0.25 mg/kg/d (N=6) | Ph 2b PMF: Bomedemstat 0.5 mg/kg/d (N=8) | Ph 2b PPV-MF: Bomedemstat 0.5 mg/kg/d (N=5) | Ph 2b PET-MF: Bomedemstat 0.5 mg/kg/d (N=11) | Ph 2b PMF: Bomedemstat 0.6 mg/kg/d (N=24) | Ph 2b PPV-MF: Bomedemstat 0.6 mg/kg/d (N=11) | Ph 2b PET-MF: Bomedemstat 0.6 mg/kg/d (N=13)
Anaemia (Blood and lymphatic system disorders) | 7 (23) | 2 (9) | 5 (34) | 2 (20) | 3 (8) | 5 (26) | 5 (5) | 3 (4) | 3 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 2 (17) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (9) | 2 (6) | 4 (19) | 7 (29) | 3 (11) | 8 (29) | 4 (11) | 6 (30) | 4 (7)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 2 (16) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 6 (8) | 4 (5) | 3 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 5 (6) | 3 (3) | 0 (0) | 4 (6) | 9 (12) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (5) | 5 (5) | 2 (2) | 3 (3) | 7 (9) | 3 (7) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (5) | 1 (3) | 2 (2) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Viral pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (7) | 3 (4) | 4 (4) | 3 (6)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blast cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 4 (5) | 0 (0) | 2 (3) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (9) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8) | 2 (2) | 3 (5) | 0 (0) | 2 (4) | 2 (2) | 5 (5) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 3 (6) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (9) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 2 (5) | 1 (1) | 2 (7) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (7) | 2 (2) | 3 (6) | 3 (3) | 0 (0) | 4 (5) | 6 (8) | 3 (4) | 5 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 2 (3)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flat affect (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 1 (1)
Phonophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0/14 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (3) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Koilonychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 2 (3) | 2 (23) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (3) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (6) | 1 (3) | 3 (4) | 2 (4) | 2 (3) | 3 (3) | 2 (2) | 2 (26) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Oedema peripheral (General disorders) | 2 (4) | 0 (0) | 1 (1) | 4 (10) | 3 (3) | 1 (1) | 4 (6) | 3 (8) | 3 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (6) | 1 (1) | 1 (2) | 1 (2)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calcium ionised decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catathrenia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperactive pharyngeal reflex (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will actively pursue publication of the results of the study in cooperation with the Lead Investigators subject to the terms and conditions of the clinical trial agreement between the Sponsor and Investigators. The Lead/Coordinating Investigator will have the right to submit for publication any results arising from the study subject to the terms and conditions of the Clinical Trial and Confidentiality Disclosure Agreements and the agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03136185/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03136185/SAP_001.pdf